CLINICAL TRIAL: NCT06945848
Title: Direct Intracranial Venous Stenting Evaluation in Patients With Idiopathic INtracranial Hypertension Under Long-term Treatment With AceTazolamidE With Inadequate Treatment Response
Brief Title: Venous Stenting Evaluation in Patients With Intracranial Hypertension Under Long-term Acetazolamide
Acronym: DIVEIINLATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL 23_0410; IDRCB (Other: 2024-A02445-42)
Record Dates: First submitted 2025-04-03; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Intracranial Hypertension (IIH)
Keywords: Intracranial hypertension; Papillary edema; Stenting; Transverse sinus vein; Chronic headache; Tinnitus
MeSH Terms: conditions — Pseudotumor Cerebri; Intracranial Hypertension; Headache Disorders; Tinnitus | interventions — Acetazolamide; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetazolamide (Active Comparator): Acetazolamide and recommended weight loss
  Interventions: Drug: Acetazolamide
- Experimental (stenting, neuro-radiological intervention) (Experimental): Stenting of the transverse sinus vein
  Interventions: Device: Stent (Tentos 4F or Precise ProRX)

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide will be maintained and weight loss will be recommended
  Other Names: Weight loss
  Arms: Acetazolamide
Device: Stent (Tentos 4F or Precise ProRX) — Transverse venous sinus will be stented by neuroradiological intervention
  Arms: Experimental (stenting, neuro-radiological intervention)

SUMMARY:
This study is aimed at patients suffering from long term intracranial hypertension (caracterized by visual loss, chronic headache and/or tinnitus), receiving acetazolamide for more than 1 year, having inadequate response to treatment (untolerable side effects or insufficient efficacy).

The goal is to evaluate if stenting of a specific vein in the brain could decrease the hypertension and improve associated symptoms. Patients will be randomly assigned in either best medical care group (recommended medication associated with weight loss) or interventional group (best medical care + stenting of the specific vein) and will undergo specific follow-up visits after 1, 3 and 12 months.

DETAILED DESCRIPTION:
The DIVE-IIN-LATE trial is a multicenter randomized controlled trial designed to evaluate whether transverse sinus stenting is more effective than best medical therapy alone for patients with idiopathic intracranial hypertension (IIH) treated with acetazolamide for more than one year. The study targets patients diagnosed with IIH with bilateral transverse sinus stenosis or unilateral stenosis of the dominant transverse sinus with a hypoplastic contralateral sinus.

Idiopathic intracranial hypertension is, in most cases, associated with narrowing of the transverse sinus vein, which may be the cause of increased intracranial blood pressure, resulting in the accumulation and increase in intracranial fluid pressure. This increased pressure is thought to be responsible for papilledema, chronic headaches, and tinnitus, among other symptoms.

Restoring a normal luminal diameter of the transverse sinus using a stent could therefore allow for the rapid restoration of normal intracranial pressures and an improvement in various symptoms.

Stent implantation in the transverse sinus is now part of standard care, but no large-scale clinical trial has formally established the superiority of the technique compared to the standard of care (drug therapy combined with weight loss). This study aims to provide evidence on the potential benefits of transverse venous sinus stenting as a treatment option for patients with idiopathic intracranial hypertension, which could significantly change the current management approach of this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old at inclusion.
2. Subject with definite diagnosis of IIH satisfying the modified Dandy criteria (A to E) ) at the time of initial diagnosis, under BMM including ACZ for more than 1 year
3. Patient with elevated intracranial pressure defined as > 25 cm H20 or 18 mmHg
4. Subject with intracranial TVS stenosis on dominant transverse sinus and hypoplastic contralateral one (or bilateral TVS stenosis) diagnosed on MRI
5. Normal MRI findings excepted intracranial TVS stenosis or IIH related abnormalities
6. Patient having received information about data collection and having signed and dated an Informed Consent Form
7. Subjects must be able to attend all scheduled visits and to comply with all trial procedures
8. Subjects must be covered by public health insurance

Exclusion Criteria:

1. Patients receiving topiramate in the previous month
2. Known contrast product, Nickel, titanium allergy
3. Exposure to an oral drug (other than ACZ), substance, or disorder that has been associated with elevation of intracranial pressure within 2 months of diagnosis (lithium, vitamin A, tetracycline and related compounds)
4. History of intracranial venous thrombosis or intracranial neoplasia
5. Fulminant decrease of visual acuity due to the IIH defined as a visual loss (of the most seriously impaired eye) of at least 3/10 (from corrected vision) within 4 weeks, in absence of any other ophthalmologic pathology and Mean Deficit of visual field superior to -10 dB
6. Optic nerve atrophy
7. Amblyopia
8. Refractive error greater ±8 sphere or more than ±3 in cylinder in either eye if there are abnormalities in funduscopy (optic disc tilt, staphyloma), previous glaucoma, other disorders causing visual loss
9. Pregnancy: if a woman is of childbearing potential a urine or serum beta HCG test is positive
10. Patient with a severe or fatal comorbidity that will likely prevent improvement or follow-up or that will render the procedure unlikely to benefit the patient.
11. Evidence of intracranial hemorrhage (subarachnoid hemorrhage (SAH), intracerebral hemorrhage (ICH), etc.)
12. Life expectancy under 6 months
13. Patients with renal failure (creatinine > 1.5 mg/dl and/or creatinine clearance < 60 mL/min, except if patient is already on hemodialysis)
14. History of previously implanted intra-cranial sinus stent
15. Previous gastric bypass surgery AAP-DGOS PHRC-N 22_0175 CHU DE MONTPELLIER Pr Costalat Vincent/Pr Ducros Anne Version n°2.2 date 25/03/2025 Page 28 sur 63
16. Contra-indication to general anesthesia
17. Contra-indication to aspirin, clopidogrel or other P2Y12 anti-aggregant
18. History of chronic obstructive pulmonary disease or other severe respiratory disease
19. History of deep vein thrombosis or pulmonary embolism
20. History of atrial fibrillation or other risks of stroke
21. Cerebral vascular lesions (arteriovenous malformation, arteriovenous fistula, aneurysms, significant stenosis of extra- or intra-cranial vessels other than the targeted venous sinus stenosis, intracranial artery dissection, etc.).
22. Anatomical anomaly of the venous sinus which would prevent safe catheterization and stenting
23. Subject who are in a dependency or employment with the sponsor or the investigator
24. Participation in another clinical trial or administration of an unapproved drug within the last 4 weeks before the screening date
25. Subject protected according to the French Public Health Code (e.g. patients under law protection, prisoners, pregnant, parturient or lactating women, and patients under guardianship/curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with normalization of intra-cranial pressure | 3 months
  Rate of patients with normalization of intra-cranial pressure (defined as ≤ 25 cm H20 or 18 mmHg)

SECONDARY OUTCOMES:
Discontinuation of Acetazolamide | 1 month
  Percentage of patients discontinuing ACZ in the stenting group without papillary edema recurrence
Discontinuation of Acetazolamide | 3 months
  Percentage of patients discontinuing ACZ in the stenting group without papillary edema recurrence
Headache | 3 and 12 months
  Change in mean HIT-6 grading scale score (patient's questionnaire containing 6 questions to evaluate the severity of headache)
Monthly headache days | 3 and 12 months
  Change in monthly headache days (within the last month) reported on patients' dairy
Tinnitus | 3 and 12 months
  Change in THI (Tinnitus Handicap Inventory) score
Visual field | 3 and 12 months
  Change in decibel of Mean Deficit visual field assessed on automated perimetry in both eyes with Humphrey Field Analyzer SITA Standard 24-2 test pattern. Each participant will have at least 2 initial visual field examinations conducted at least 30 minutes apart. The 2 Perimetric Mean Deviation (PMD) measurements will be averaged.
Visual acuity | 3 and 12 months
  Change of visual acuity score evaluated on ETDRS (far vision) at 4 meters and reproducible lighting using the best optical correction
Visual acuity | 3 and 12 months
  Change of visual acuity score evaluated on Parinaud scale (near vision) using the best optical correction
Papilledema | 3 and 12 months
  Change of papilledema assessed on Frisen score on OCT
Papilledema | 3 and 12 months
  Change of papilledema assessed on RNFL on OCT
Patient's autonomy | 3 and 12 months
  Change in quality of life assessed on EQ5D questionnaire
Patient's cognition | 3 and 12 months
  Change in Montreal Cognitive Assessment (MoCA)
Cognition | 3 and 12 months
  Change in Trail Making Test (TMT)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent COSTALAT, MD, PhD, Study Director — University hospital of Montpellier, FRANCE
Locations (3):
- France (3):
  - CHU de Montpellier Hôpital Gui de Chauliac, Montpellier
  - CHU de Reims, Reims
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No